CLINICAL TRIAL: NCT05830526
Title: Nursing Students' Evaluation of the Preoperative Period ERAS Protocol: An Example of an Escape Room
Brief Title: Example of Escape Room in Nursing Student Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Refiye Akpolat, Assistant Proffesor, Kocaeli University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 112345678
Record Dates: First submitted 2023-03-23; First posted 2023-04-26 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Education, Nursing
Keywords: Escape Room; İnnovative Learn; Nursing Students; educational game

STUDY DESIGN:
Masking Description: Groups of 5 people were formed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Escape Room (Other): All of the participants were trained in the escape room.
  Interventions: Other: Escape Room

INTERVENTIONS:
Other: Escape Room — The next day, 56 students, who agreed to participate in the study, were divided into groups of 5, and they had to fill out a 10-question test, which includes the stages of the ERAS Protocol preoperative period, within the scope of the pre-test. A simulation room for students has been set up as an escape room. At the briefing on the theme of the escape room, it was explained that they would have 10 minutes to complete six missions using the clues given to them.
  The 6 stations created in the room were numerically numbered from 1 to 6. There were question/answer cards at each station and a clue on the back of the correct answer card to reach the next station. The first clue was given by the observer who made the information in the information room.The student who could not get out of the room within 10 minutes was considered as unable to leave the escape room.

SUMMARY:
Game-based learning is gaining increasing attention to meet the evolving needs of today's nursing students and the demand for 21st century skills in modern healthcare. After the COVID-19 pandemic, the need for innovative learning methods has increased in the process of transferring the theoretical knowledge of nursing students into practice. It can improve learning outcomes while enhancing learning experiences by encouraging participation and motivation. Different teaching methods are used during the teaching of the course they take to nursing students. Game-based learning, which is one of them, is used to increase the motivation of students and to contribute to the acquisition and evaluation of knowledge and skills. Escape room is one of the methods used in this area.

The integration of innovative strategies into teaching and learning in higher education, such as escape room games as a learning method, has been reported to increase the acquisition of key professional competences, including communication, teamwork, and critical thinking. Within the scope of the innovative learning method, it is aimed that nursing students correctly evaluate the preoperative steps of the Enhanced Recovery After Surgery protocol in the escape room so that they can use the theoretical knowledge they have received in this study in practice.

DETAILED DESCRIPTION:
Data Collection Tools Pretest-Posttest: The content of the test, which was prepared by a specialist in the field of surgical nursing, consisted of 10 multiple-choice questions belonging to the preoperative steps of the Enhanced Recovery After Surgery protocol. Students completed the test before entering the escape room and immediately after leaving the room. The maximum score from the test was 100.

After leaving the escape room, the students were questioned about their satisfaction with the game training.Theoretical information including Enhanced Recovery After Surgery (ERAS) protocol was given to the students 1 day before the application. The next day, 56 students, who agreed to participate in the study, were divided into groups of 5, and they had to fill out a 10-question test, which includes the stages of the ERAS Protocol preoperative period, within the scope of the pre-test.

A simulation room for students has been set up as an escape room. The room was likened to a patient room in a clinic. Before entering the escape room, students were read the demographic and medical information of a patient who will undergo gynecological surgery in the information room next to the simulated patient room. Later, in the briefing about the escape room theme, it was announced that they would have 10 minutes to complete six missions using the clues given to them. Students who could not leave the room within 10 minutes were considered unsuccessful.

ELIGIBILITY:
Inclusion Criteria:

* Having received Enhanced Recovery After Surgery protocol training
* Being a 3rd Year Nursing Student
* Voluntary participation in the study

Exclusion Criteria:

* Those who did not receive Enhanced Recovery After Surgery protocol training
* Non 3rd Year Nursing Student
* unwilling to participate in the study

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Escape from the educational game room | 10 minutes
  93 students from the 3rd grade nursing department formed the universe of the project. The sample consisted of 56 students who agreed to participate in the research. The students were given theoretical training on the preoperative steps of the Enhanced Recovery After Surgery Protocol. One day later, a simulation room was set up where they would repeat the theoretical training they received in practice. In the room, which was adapted as a patient room, the stations where the questions related to each step of the theoretical education given to the students were determined. The 6 stations created in the room were numerically numbered from 1 to 6. After the students gave the correct answer to the questions they found at each station, they went to the next station. It was announced that they would have 10 minutes to complete all stations. Students who completed the task within 10 minutes were considered to have exited the escape room.
Effect of escape room game on knowledge level | 2 days
  The questions about the theoretical training of the ERAS protocol, which they had received the day before, were administered to the students as a pretest-posttest before they were admitted to the game room and after they left the game room. With the escape room game application, the recall of theoretical knowledge and the increase in the level of knowledge compared to the pretest were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Refiye Akpolat, Principal Investigator — Kocaeli Healt and Tecnology University
Locations (1):
- Kocaeli Healt and Tecnology University, Kocaeli, Başiskele, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No